CLINICAL TRIAL: NCT01669733
Title: The Effects of Perioperative Music Therapy on Women Undergoing Breast Biopsy Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE5112
Record Dates: First submitted 2012-08-16; First posted 2012-08-21 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Abnormal Breast Tissue
Keywords: Breast Surgery; Breast Biopsy; Music Therapy
MeSH Terms: interventions — Music Therapy; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Live/Recorded Music Group (Experimental): The music therapist will prepare a preferred song to be performed live in the preoperative room. Subjects in the live music group will listen to recorded music intraoperatively.
  Interventions: Other: Music
- Recorded Music Group (Experimental): Recorded music group will be given an iPod and headphones and will listen to a recorded version of a preferred song.
  Interventions: Other: Music
- No Music (Standard of care) (Active Comparator): The control group will receive standard of care and no music.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Music — Recorded or live music will be played prior to surgery in the preoperative room. Subjects in the live music group and subjects in the recorded music group will listen to recorded music intraoperatively. An ipod with headphones will be given to the subject when she is being prepared to move to the operating room. The board certified music therapist will initiate recorded music (harp selections). Recorded music will be relaxing harp selections. The board certified music therapist will accompany the subject to the operating room and assure volume levels and electronic equipment function properly.
  Other Names: Recorded Music; Live Music
  Arms: Live/Recorded Music Group; Recorded Music Group
Other: Standard of Care — The control group subjects will receive standard anesthesia, nursing and surgical care.
  Arms: No Music (Standard of care)

SUMMARY:
The purpose of this research is to study the effect music has on women undergoing surgical breast biopsy. Through the facilitation of live and/or recorded music listening, we will examine the perception of patient anxiety, the total amount of propofol required to obtain a BIS reading of 70, and recovery time in the PACU. We will also collect data and evaluate the effect of live and/or recorded music on patient satisfaction. It is hypothesized that:

1. Patients in the live and recorded music groups will experience less anxiety than the non-music (standard care) group.
2. Patients in the live and recorded music groups will experience a reduction in the amount of anesthesia needed to reach a state of moderate sedation compared to the non-music (standard care) group.

DETAILED DESCRIPTION:
Music therapy's effect on anxiety in Preoperative.(live vs. recorded):

If the patient is randomly selected to the live music group, the music therapist will prepare a preferred song to be performed live in the preoperative room. If the patient is randomly selected for the recorded music group, she will be given an iPod and headphones and will listen to a recorded version of her preferred song. If the patient is randomly selected for the control group, she will receive standard care and no music. Pre/posttests will be given using a Global Anxiety Visual Analog Scale (GA-VAS).

Music therapy's effect on propofol requirements intraoperatively:

Subjects in the live music group and subjects in the recorded music group will listen to recorded music intraoperatively. All subjects will receive equal amounts of fentanyl and versed. Subjects will receive fentanyl in the amount of 1 microgram per kilogram and versed (midazolam) in the amount of 0.02 milligrams per kilogram from the nurse anesthetist. An ipod with headphones will be given to the subject when she is being prepared to move to the operating room. The board certified music therapist will initiate recorded music (harp selections). Recorded music will be relaxing harp selections. The board certified music therapist will accompany the subject to the operating room and assure volume levels and electronic equipment function properly.

Anesthesia personnel will apply BIS monitor before propofol administration. Anesthesia personnel will titrate propofol to obtain BIS reading of 70 or lower and record the propofol in micrograms per kilogram per minute, infusing at that point. Signal Quality Index (SQI) will be recorded when the BIS reaches 70 to give credibility to the BIS monitor. SQI is a measure of the signal quality for the EEG channel source and is calculated based on impedance data, artifact, and other variables. The total amount of propofol for the case will be recorded as total milligrams received. Anesthesia personnel will record Observer's Assessment of the Alertness/Sedation (OAA/S) when BIS monitor reaches 70 or below as incidental data point. A score of 3 on OAA/S indicates that the patient responds only after mild prodding and shaking. OAA/S will be compared to BIS reading.

Time in PACU and Patient Satisfaction:

Recorded music will continue playing until the subject has met discharge criteria according to University Hospital's policy and procedure. The amount of time between when the patient leaves the operating room and meets discharge criteria (determined by nurse) will be recorded. Patient satisfaction will be recorded using a Likert scale: 7= highly satisfied; 1=not at all satisfied after the subject has met her discharge criteria.

Controls: The control group subjects will receive standard anesthesia, nursing and surgical care. All rating procedures will be the same. Controls will wear noise reducing headphones. The music therapist will not accompany control patients following surgery. When the trial is complete, the music therapist will offer the control subject a CD of the recorded music once she has met discharge criteria and all data is recorded. This will occur for the sake of ethics.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who will undergo surgical breast biopsy under monitored anesthesia care
* English speaking women
* >18 years
* ASA classification of I (no systematic disease) or II (mild to moderate disease who are medically stable) or III (severe systematic disease, not incapacitating)

Exclusion Criteria:

* Patients with profound mental illness
* with developmental disability
* with significant hearing loss where music would not be heard from headphones
* currently taking narcotics

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2012-08; Primary Completion 2014-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
The cumulative intra-operative dose of propofol(mg) given to each patient | at the time of surgery
  The primary outcome for this study will be the amount of propofol administered intra-operatively. Each of the groups receiving music pre-operatively and/or peri-operatively will be compared to the control (no music) group. Anesthesia personnel will apply BIS (Bispectral Index Monitor) monitor before propofol administration. Anesthesia personnel will titrate propofol to obtain BIS reading of 70 or lower and record the propofol in micrograms per kilogram per minute, infusing at that point. The total amount of propofol for the case will be recorded as total milligrams received.
Change in anxiety levels | Pr- and post- music therapy prior to surgery
  Pre/posttests will be given using a Global Anxiety Visual Analog Scale (GA-VAS). A pretest will be given in the preoperative area before intervention and a posttest will be given after the live song, the recorded song, or five minutes of standard care has occurred. The investigators will measure the subject's marking (vertical line) on the GA-VAS from the left side of the GA-VAS to the subject's line using millimeters on a ruler.

SECONDARY OUTCOMES:
Amount of time in the PACU (post-anesthesia care unit) | at time of discharge from PACU
  Amount of time between when the patient leaves the operating room and meets discharge criteria (determined by nurse) using a clock.
Patient satisfaction to music therapy | at the time of PACU discharge
  Qualitative data will be taken on the subject's subjective comments regarding their thoughts about their surgical experience using a 1-10 Likert Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Deforia Lane, PhD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States